CLINICAL TRIAL: NCT05410691
Title: Handheld Ultrasound-guided Cannulation of Difficult Haemodialysis Arteriovenous Access by Renal Nurses - A Randomised Controlled Trial
Brief Title: Handheld Ultrasound-guided Cannulation of Difficult Haemodialysis Arteriovenous Access by Renal Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Allen Liu Yan Lun, Senior Consultant, National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEG2022
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Hemodialysis Complication; Dialysis; Complications; Vascular Access Site Haematoma; Vascular Access Complication; Dialysis Access Malfunction; Fistula; Graft Av
Keywords: haemodialysis; dialysis; arteriovenous fistula; arteriovenous graft; ultrasound; vascular access
MeSH Terms: conditions — Fistula; Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): AVF/AVG cannulation by renal nurses in standardised manner
- ultrasound guided (Active Comparator): AVF/AVG cannulation by renal nurses by handheld US device
  Interventions: Device: Handheld US device

INTERVENTIONS:
Device: Handheld US device — Handheld US-guided AVF/AVG cannulation
  Arms: ultrasound guided

SUMMARY:
Cannulation of complex arteriovenous fistula (AVF) or graft (AVG) is a challenge to renal nurses. Ultrasound (US) guidance on central and peripheral venous access visualisation has been widely adopted in nephrology and shown to reduce complications of vascular interventions. With broader adoption of handheld US devices in clinical services, renal nurses could acquire this point-of-care technique to increase the successful cannulation rate while facilitating confidence build-up during training and practice. We aim to evaluate the use of handheld US on difficult AVF/AVG cannulation in a hospital-based dialysis unit.

DETAILED DESCRIPTION:
We conducted a prospective randomised controlled study from January 2021 to January 2022. Ten renal nurses were trained by an interventional nephrologist before patient recruitment and had completed a pre- and post-training questionnaire on their confidence level. Fifty haemodialysis patients with complex AVF were randomised to US-guided or conventional cannulation. The total time spent on cannulation and patients' pain scores were also collected.

ELIGIBILITY:
Inclusion Criteria:

1. First-time cannulation, 2. Post-angioplasty or thrombectomy, 3. Partial stenosis confirmed with imaging or by vascular surgeons/interventional radiologists, 4. Failed cannulation by dialysis nurses at community centres, 5. Bruises or haematoma around AVF/AVG, 6. Presence of clots in AVF/AVG and 7. Deep-seated access by physical examination.

Exclusion Criteria:

complex access with a high risk of complications (calibre ≤0.4cm or vessels ≥0.8cm in depth from skin)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
percentage of successful cannulation | from skin contact to actual start of dialysis

SECONDARY OUTCOMES:
pre-cannulation assessment time | from patient physical contact to the time before needling thru skin
  time taken to assess the AVF/AVG with either US or clinical examination before cannulation
cannulation time | skin contact by needle to succesful aspiration of blood from needle
patients' pain score | needle to skin to end of dialysis session
  10cm visual analogue scale
complications | from skin contact to actual start of dialysis
  need for a temporary central venous catheter, single-needle dialysis, or infiltration (e.g. haematoma) that hastened the use of AVF/AVG for the same dialysis session

CONTACTS AND LOCATIONS:
Overall Officials: Shune Chen, Principal Investigator — NHG, Khoo Teck Puat Hospital
Locations (1):
- Allen Liu, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No